CLINICAL TRIAL: NCT02655120
Title: Evaluation of the Efficiency of Autologous Bone Marrow no Concentrated to Associate at BMP7 Treatment of Necrosis of the Femoral Head of the Adult
Brief Title: Autologous Bone Marrow and BMP7 Treatment in the Necrosis in the Femoral Head of the Adult
Acronym: BMP7
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: stopping the marketing of BMP7
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-0503; TC 183 (Other: therapy cellulaire number, ANSM)
Record Dates: First submitted 2014-11-12; First posted 2016-01-13 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Aseptic Necrosis of Femur Head
Keywords: Femoral head necrosis; Autologous Bone Marrow; BMP7
MeSH Terms: conditions — Femur Head Necrosis | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bone Marrow +BMP7 (Experimental): The drilling is completed by a joint supply of autologous marrow unconcentrated and recombinant BMP7 (OP1)
  Interventions: Biological: Bone Marrow +BMP7
- Drilling (Placebo Comparator): Group I: a simple drill is practiced
  Interventions: Procedure: Drilling

INTERVENTIONS:
Procedure: Drilling
  Arms: Drilling
Biological: Bone Marrow +BMP7
  Arms: Bone Marrow +BMP7

SUMMARY:
The main objective of the study is to evaluate the effectiveness of the injection of bone marrow unconcentrated more R BMP 7 to repair necrosis of the femoral head with stage I-III classification FICAT.

DETAILED DESCRIPTION:
Rationale and Objectives Epiphyseal necrosis are common in young adults (2000 new cases per year in the Nord Pas -de- Calais region) resulting in severe functional impairment and disability . Drilling is the procedure most simple, but its effectiveness and safety are discussed ( fracture risk , long discharge period , success rates below 50 % until stage III). However, it can be optimized in two ways: 1) reducing morbidity and discharge period by reducing the diameter of the channel and percutaneous achievement , 2 ) increase efficiency , including coverage contribution of stem cells and osteogenic hormone . The purpose of this study is to test the effectiveness of the contribution of these elements to the healing necrosis .

Material, Method, and primary endpoint This is a prospective multicenter clinical trial randomized double-blind . The effect of addition of autologous bone marrow stem cells and BMP7 on healing necrosis is assessed by magnetic resonance imaging ( NMRI ) and is the primary endpoint . Patients are randomly assigned to two arms : 1 ) Group I: a simple drilling is practiced , 2 ) Group II : the drilling is completed by a joint supply of autologous marrow unconcentrated and recombinant BMP7 ( OP1 ) . Necrosis of the femoral head with stage I to III are retained Ficat (only stage III with a recess of less than 3 mm are used , corresponding I-III according to Steinberg ) . Forty patients are included in each arm . A IRMN practiced preoperatively and at 6 months and 2 years. Clinical evaluation will be continued up to 5 years in testing the survival rate ( criterion censorship = recovery by hip ) Expected results and possible implications In terms of radiological stabilization ( NMRI ) the effectiveness of single drilling necrosis stage I to III Ficat is 60 % ( non- stabilization or worsening of size). The hypothesis tested is a gain stabilization ( and / or recovery) of 20 % . The clinical efficacy of single drilling necrosis stage I to III Ficat is estimated at 50 % (50% recovery by prosthesis in 5 years) . The assumption is a 20% improvement in the rate of success of the intervention . Reducing morbidity due to technical modifications has been previously tested. If the assumption of success is reached, the indications of drilling could be reinforced especially for patients with multiple visceral defects usually supported on the websites of University Hospital of Lille and Amiens and CH Roubaix ( organ transplant or tissue , ethyl , .. ) .

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 18 and 60 years male or female.
* Necrosis of the femoral head stage I to III FICAT (stage III with depression of less than 3 mm)
* Nontraumatic osteonecrosis
* Patient can undergo general anesthesia or locoregional
* Having given his consent
* Able to understand the constraints of the study

Exclusion Criteria:

* Refusing to participate in the study
* Active infection at the site
* Cancer changing
* Pregnancy
* Necrosis posttraumatic
* Having already undergone surgery on the surgical site
* Contraindication to the practice of NMRI
* Contraindication to the use of OP1 (BMP7): collagen, arthritis, scleroderma, lupus
* Patient participating in another ongoing study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2005-03; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Necrosis volume | 24 months
  Varying the volume of necrosis in MRI, student test comparing the mean (independent samples).

SECONDARY OUTCOMES:
Merle d'aubigné hip score | 6 and 24 months
  variation of functional score, according to the two groups, by ANOVA repeated measures
Measurement of radiographic stage variation between pre-operative and 24 months radiographies using concentric circles of Möse | 24 months
Comparison of hip survival by measuring the number of revisions for hip replacement in the 2 groups | 60 months
  Hip survival (= no revision for hip replacement) will be assessed using Kaplan-Meier curves and Logrank test.

CONTACTS AND LOCATIONS:
Overall Officials: Henri Migaud, MD, PhD, Study Chair — University Hospital, Lille
Locations (1):
- CHRU de LILLE - service d'orthopédie C, Lille, France